CLINICAL TRIAL: NCT00513721
Title: Do Positive Lateral Biopsy Cores on TRUS Directed Biopsies Predict Capsular Penetration and Positive Surgical Margins?
Brief Title: Retrospective Study of Positive Biopsy Specimens on Patients Undergoing a Prostatectomy
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Kenneth Peters, William Beaumont Hospital
Other Study IDs: E2007-087
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Prostate Cancer
Keywords: prostate; prostate cancer; surgical margins; gleason score; positive lateral biopsies
MeSH Terms: conditions — Prostatic Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- III: Prostate specimens with positive surgical margins.

SUMMARY:
This is a review of prostate biopsy specimens which show capsular penetration or positive surgical margins. Patients had surgery performed at William Beaumont Hospital-Royal Oak, Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Males having undergone surgery for prostate cancer at William Beaumont Hospital-Royal Oak, Michigan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males having undergone surgery for prostate cancer at William Beaumont Hospital-Royal Oak, Michigan
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Eliya, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States